CLINICAL TRIAL: NCT02359110
Title: Administration of Pre-Operative Gabapentin to Patients Undergoing Laparoscopy: A Prospective Double-blinded, Placebo Controlled Randomized Study
Brief Title: Administration of Pre-Operative Gabapentin to Patients Undergoing Laparoscopy
Acronym: Gabapentin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Timothy A Deimling, Principal Investigator; Minimally Invasive Gyn Surgery Fellow, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1183
Record Dates: First submitted 2015-02-04; First posted 2015-02-09 (Estimated); Results first posted 2018-03-12 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Postoperative Pain
Keywords: laparoscopy; postoperative pain; gynecology; gabapentin
MeSH Terms: conditions — Pain, Postoperative | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug 1 (Experimental): Patients will receive Gabapentin 300mg tab less than 1 hour before surgery.
  Interventions: Drug: Gabapentin
- Drug 2 (Placebo Comparator): Patients will receive Methylcellulose based placebo tab less than 1 hour before surgery.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Gabapentin — Patients will receive Gabapentin 300mg tab less than 1 hour before surgery.
  Other Names: Neurontin; 78309289
  Arms: Drug 1
Other: Placebo — Patient will receive placebo tab less than 1 hour before surgery
  Arms: Drug 2

SUMMARY:
The purpose of this study is to prospectively determine the influence of immediate pre-operative gabapentin administration on acute postoperative pain. The investigators hypothesize that immediate post-operative pain will be improved with pre-operative administration of gabapentin.

DETAILED DESCRIPTION:
The purpose of this study is to prospectively determine the influence of immediate pre-operative gabapentin administration on acute postoperative pain. We hypothesize that immediate post-operative pain will be improved with pre-operative administration of gabapentin.

We plan to conduct a prospective randomized trial to assess the effect of a single immediate pre-operative dose of gabapentin 300mg on immediate post-operative pain in patients undergoing laparoscopy for gynecologic indications. This concept has been studied in patients undergoing abdominal hysterectomy. We aim to study the effect on patients undergoing laparoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be female and planning to have a laparoscopic or robotic assisted procedure for benign gynecologic indications.
2. Patients must be treated in the department of Obstetrics and Gynecology in the division of Minimally Invasive Gynecologic Surgery.
3. The patient must be in the age range of 18-80 years, in general good health and able to comply with study procedures.

Exclusion Criteria:

1. Male patients will be excluded from this study.
2. Patients under 18 years old will be excluded from this study.
3. Pregnant patients. All patients will have a routine pre-operative urine HCG to exclude pregnancy.
4. Patients having abdominal, vaginal or hysteroscopic procedures
5. Allergy to gabapentin
6. Chronic use of gabapentin (greater than 6 months)

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2015-06; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Walker JL, Piedmonte MR, Spirtos NM, Eisenkop SM, Schlaerth JB, Mannel RS, Spiegel G, Barakat R, Pearl ML, Sharma SK. Laparoscopy compared with laparotomy for comprehensive surgical staging of uterine cancer: Gynecologic Oncology Group Study LAP2. J Clin Oncol. 2009 Nov 10;27(32):5331-6. doi: 10.1200/JCO.2009.22.3248. Epub 2009 Oct 5. PMID 19805679
- [Background] Manwaring JM, Readman E, Maher PJ. The effect of heated humidified carbon dioxide on postoperative pain, core temperature, and recovery times in patients having laparoscopic surgery: a randomized controlled trial. J Minim Invasive Gynecol. 2008 Mar-Apr;15(2):161-5. doi: 10.1016/j.jmig.2007.09.007. PMID 18312984
- [Background] Ott DE, Reich H, Love B, McCorvey R, Toledo A, Liu CY, Syed R, Kumar K. Reduction of laparoscopic-induced hypothermia, postoperative pain and recovery room length of stay by pre-conditioning gas with the Insuflow device: a prospective randomized controlled multi-center study. JSLS. 1998 Oct-Dec;2(4):321-9. PMID 10036122
- [Background] Sills GJ. The mechanisms of action of gabapentin and pregabalin. Curr Opin Pharmacol. 2006 Feb;6(1):108-13. doi: 10.1016/j.coph.2005.11.003. Epub 2005 Dec 22. PMID 16376147
- [Background] Hartrick CT, Kovan JP, Shapiro S. The numeric rating scale for clinical pain measurement: a ratio measure? Pain Pract. 2003 Dec;3(4):310-6. doi: 10.1111/j.1530-7085.2003.03034.x. PMID 17166126
- [Background] Clarke H, Bonin RP, Orser BA, Englesakis M, Wijeysundera DN, Katz J. The prevention of chronic postsurgical pain using gabapentin and pregabalin: a combined systematic review and meta-analysis. Anesth Analg. 2012 Aug;115(2):428-42. doi: 10.1213/ANE.0b013e318249d36e. Epub 2012 Mar 13. PMID 22415535
- [Background] Alayed N, Alghanaim N, Tan X, Tulandi T. Preemptive use of gabapentin in abdominal hysterectomy: a systematic review and meta-analysis. Obstet Gynecol. 2014 Jun;123(6):1221-1229. doi: 10.1097/AOG.0000000000000289. PMID 24807337
- [Background] Alkhamesi NA, Peck DH, Lomax D, Darzi AW. Intraperitoneal aerosolization of bupivacaine reduces postoperative pain in laparoscopic surgery: a randomized prospective controlled double-blinded clinical trial. Surg Endosc. 2007 Apr;21(4):602-6. doi: 10.1007/s00464-006-9087-6. Epub 2006 Dec 16. PMID 17180268
- [Background] Nutthachote P, Sirayapiwat P, Wisawasukmongchol W, Charuluxananan S. A randomized, double-blind, placebo-controlled trial of oral pregabalin for relief of shoulder pain after laparoscopic gynecologic surgery. J Minim Invasive Gynecol. 2014 Jul-Aug;21(4):669-73. doi: 10.1016/j.jmig.2014.01.018. Epub 2014 Jan 25. PMID 24473153

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 125 patients consented to the study, but 13 did not undergo surgery or rescheduled.
Pre-assignment Details: A total of 112 patients were enrolled, but 3 did not receive study drug.
Groups:
- Placebo: Patients will receive Methylcellulose based placebo tab less than 1 hour before surgery.
Period: Overall Study
Arm/Group | Gabapentin | Placebo
Started | 55 | 54
Completed | 55 | 54
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin | Placebo | Total
Number analyzed (Participants) | 55 | 54 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (9.8) | 39.5 (9.4) | 39.9 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 54 | 109
  Male | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m2] | 29.5 (7.2) | 30.0 (7.7) | 29.8 (7.4)

OUTCOME MEASURES:

1. Primary Outcome: NRS (Numerical Rating Scale)
Description: The NRS is a numerical scale ranging from 0-10 implemented with adults. Having no pain is rated as a 0 and the worst pain the patient could tolerate is rated as a 10.
Time Frame: 2-8 hours
Population: Our analysis uses all available data. Some participants were not in house for the full 8 hours of collection, others did not complete NRS at the respective time point. Therefore the number at each time point differs from the overall number of participants.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 55 | 54
units on a scale
  Hour 2: number analyzed (Participants) | 46 | 49
  Hour 2 | 3.5 [2.6 to 4.5] | 3.4 [2.5 to 4.4]
  Hour 4: number analyzed (Participants) | 28 | 25
  Hour 4 | 5.4 [4.3 to 6.5] | 5.5 [4.3 to 6.7]
  Hour 6: number analyzed (Participants) | 30 | 19
  Hour 6 | 5.3 [4.2 to 6.5] | 5.8 [4.4 to 7.1]
  Hour 8: number analyzed (Participants) | 23 | 17
  Hour 8 | 5.7 [4.3 to 7.2] | 5.1 [3.4 to 6.8]
Statistical Analysis 1: Comparison: Gabapentin vs Placebo; Hour 2 Analysis; Test type: Superiority; p = 0.89, Mixed Models Analysis; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-1.2 to 1.3]
Statistical Analysis 2: Comparison: Gabapentin vs Placebo; Hour 4 Analysis; Test type: Superiority; p = 0.94, Mixed Models Analysis; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-1.6 to 1.5]
Statistical Analysis 3: Comparison: Gabapentin vs Placebo; Hour 6 Analysis; Test type: Superiority; p = 0.64, Mixed Models Analysis; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-2.2 to 1.3]
Statistical Analysis 4: Comparison: Gabapentin vs Placebo; Hour 8 Analysis; Test type: Superiority; p = 0.59, Mixed Models Analysis; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-1.6 to 2.8]

2. Secondary Outcome: VAS (Visual Analog Scale)
Description: The VAS is scored using a horizontal line 100mm in length. The scale is anchored by "no pain" (score of 0) and "worst pain" (score of 100).
Time Frame: 2 -6 hours
Population: Our analysis uses all available data. Some participants were not in house for the full 6 hours of collection, others did not complete VAS at the respective time point. Therefore the number at each time point differs from the overall number of participants.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 55 | 54
units on a scale
  Hour 2: number analyzed (Participants) | 31 | 32
  Hour 2 | 37.8 [28.9 to 46.6] | 33.9 [25.3 to 42.6]
  Hour 6: number analyzed (Participants) | 25 | 24
  Hour 6 | 38.7 [28.6 to 48.7] | 36.9 [26.9 to 46.9]
Statistical Analysis 1: Comparison: Gabapentin vs Placebo; Hour 2 Analysis; Test type: Superiority; p = 0.52, Mixed Models Analysis; Mean Difference (Final Values) = 3.8, 95% CI 2-sided [-8.1 to 15.8]
Statistical Analysis 2: Comparison: Gabapentin vs Placebo; Hour 6 Analysis; Test type: Superiority; p = 0.80, Mixed Models Analysis; Mean Difference (Final Values) = 1.7, 95% CI 2-sided [-11.9 to 15.3]

3. Secondary Outcome: Total Morphine Consumption
Time Frame: 12 hours post-operatively
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 55 | 54
mg | 14.3 (12.6) | 14.7 (12.3)
Statistical Analysis 1: Comparison: Gabapentin vs Placebo; Test type: Superiority; p = 0.88, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Gabapentin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/54
Other Adverse Events (participants affected / at risk) | 0/55 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No